CLINICAL TRIAL: NCT01174667
Title: Effect of Fascial Release on Connective Tissue Structure in Human Subjects With Chronic Low Back Pain as Determined by Ultrasound Imaging: a Randomized Controlled Trial
Brief Title: Massage of the Low Back Muscles Assessed With Ultrasound Scanning
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anglo-European College of Chiropractic (Other)
Responsible Party: Hugh Gemmell Principal Lecturer, Anglo-European College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AECC 290710
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-07

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial pain; Trigger points
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascial massage (Experimental): A specific type of fascial massage to release restricted lumbodorsal fascia.
  Interventions: Procedure: Specific massage for fascial release
- No treatment control (No Intervention): Patient will rest quietly without receiving any instruction.
  Interventions: Other: Quiet non-instructed rest for 3 minutes

INTERVENTIONS:
Procedure: Specific massage for fascial release — Patient will receive a 3 minute massage to reduce restrictions in the lumbodorsal fascia.
  Other Names: Superficial fascial release
  Arms: Fascial massage
Other: Quiet non-instructed rest for 3 minutes — Patient will lay quietly without any instructions on how to relax.
  Other Names: Uninstructed rest
  Arms: No treatment control

SUMMARY:
The aim of the study is to use diagnostic ultrasound to compare the thickness of soft tissues in the low back in a group of patients with chronic low back pain treated with massage to a control group of non-treated patients.

It is hypothesized that on average, soft tissue thickness in the lumbar region will change in the group receiving massage compared to the control group.

DETAILED DESCRIPTION:
A specialized form of massage designed to reduce fascial restrictions will be compared to a no-treatment control group based on a change in thickness of the lumbodorsal fascia as determined by ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic low back pain far at least 3 months
* Able to read and write English
* Between 18-64 years of age

Exclusion Criteria:

* Prior lumbar surgery
* Infected or broken skin over the lumbodorsal fascia
* Major structural spinal deformity
* Specific cause of low back pain, such as tumor, infection, fracture
* Bleeding disorders or use of anticoagulant medications
* Pregnancy
* Litigation for low back pain
* Systemic infection

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Thickness of lumbodorsal fascia determined by ultrasound imaging | An average of 5 minutes from the the end of first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Gemmell, DC, EdD, Principal Investigator — Anglo-European College of Chiropractic